CLINICAL TRIAL: NCT04777812
Title: Pancreatitis - Microbiome As Predictor of Severity
Acronym: P-MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Collaborators: Department of Medicine II, University Hospital Rostock (Unknown); Medical Department II, Division of Gastroenterology, University Hospital of Leipzig (Unknown); Department of Medicine II, University Hospital, LMU Munich (Unknown); Department of Medicine I, University Hospital of Halle (Unknown); Department of Medicine A, University Medicine Greifswald (Unknown); Department of Medicine II, University Hospital rechts der Isar, Technical University Munich (Unknown); Department of Medical Bioinformatics, University Medical Center Göttingen (Unknown); Department if Medical Statistics, University Medical Center Göttingen (Unknown)
Responsible Party: Principal Investigator, Albrecht Neesse, Prof. Dr. Dr., University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-MAPS_02794
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rectal and buccal swabs — The oral and intestinal flora is collected from buccal and rectal swabs.

SUMMARY:
This study is a multicentric prospective study initiated and coordinated from the University Medical Centre Goettingen. The study aims to evaluate the orointestinal microbiome as a potential biomarker for the course, severity and outcome of patients with acute pancreatitis.

DETAILED DESCRIPTION:
This prospective translational study aims to evaluate the orointestinal microbiome as a potential biomarker for the course, severity and outcome of patients with acute pancreatitis. From each patient one buccal and rectal swab is collected within 72 h after hospital admission. Microbial composition will be determined by 16S and metagenomics Oxford Nanopore Sequencing (ONT) and correlated with the revised Atlanta classification as the primary endpoint. Secondary endpoints are the correlation of microbiome signatures with the length of hospital stay, numbers of interventions and mortality. To this end, alpha and beta diversity of microbiota are determined and compared between mild, moderately severe and severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute pancreatitis (2 out of 3 following diagnostic criteria: lipase >3x of upper limit, abdominal pain, and imaging modalities (computed tomography, magnetic resonance imaging or ultrasound).

< 72 hours after hospital admission.

Exclusion Criteria:

Pregnant women Patients < 18 years; Patients who are incapable of giving consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Revised Atlanta classification I-III | up to 8 weeks
  Microbial composition (alpha and beta-diversity) will be correlated with the revised Atlanta classification.

SECONDARY OUTCOMES:
Length of hospital stay | up to 12 months
  days in hospital during initial admission
Numbers of interventions (surgical and endoscopical) | up to 12 months
  number of percutaneous drainages, number of EUS-guided interventions of infected necrotic or acute collections, type of drainages (plastic versus lumen apposing metal stents), number of open surgical interventions
Mortality | up to 12 months
  in hospital mortality during initial admission (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammer-Herrmenau C, Pfisterer N, Weingarten MF, Neesse A. The microbiome in pancreatic diseases: Recent advances and future perspectives. United European Gastroenterol J. 2020 Oct;8(8):878-885. doi: 10.1177/2050640620944720. Epub 2020 Jul 23. PMID 32703080
- [Background] Ammer-Herrmenau C, Antweiler KL, Asendorf T, Beyer G, Buchholz SM, Cameron S, Capurso G, Damm M, Dang L, Frost F, Gomes A, Hamm J, Henker R, Hoffmeister A, Meinhardt C, Nawacki L, Nunes V, Panyko A, Pardo C, Phillip V, Pukitis A, Rasch S, Riekstina D, Rinja E, Ruiz-Rebollo ML, Sirtl S, Weingarten M, Sandru V, Woitalla J, Ellenrieder V, Neesse A. Gut microbiota predicts severity and reveals novel metabolic signatures in acute pancreatitis. Gut. 2024 Feb 23;73(3):485-495. doi: 10.1136/gutjnl-2023-330987. PMID 38129103
- [Derived] Ammer-Herrmenau C, Meier R, Antweiler KL, Asendorf T, Cameron S, Capurso G, Damm M, Dang L, Frost F, Hamm J, Hoffmeister A, Kocheva Y, Meinhardt C, Nawacki L, Nunes V, Panyko A, Ruiz-Rebollo ML, Florez-Pardo C, Phillip V, Pukitis A, Vaselane D, Rinja E, Sandru V, Schaefer A, Scholz R, Seelig J, Sirtl S, Ellenrieder V, Neesse A. Gut microbiota predict development of postdischarge diabetes mellitus in acute pancreatitis. Gut. 2026 Jan 8;75(2):316-325. doi: 10.1136/gutjnl-2025-336715. PMID 41298102
- [Derived] Ammer-Herrmenau C, Asendorf T, Beyer G, Buchholz SM, Cameron S, Damm M, Frost F, Henker R, Jaster R, Phillip V, Placzek M, Ratei C, Sirtl S, van den Berg T, Weingarten MJ, Woitalla J, Mayerle J, Ellenrieder V, Neesse A. Study protocol P-MAPS: microbiome as predictor of severity in acute pancreatitis-a prospective multicentre translational study. BMC Gastroenterol. 2021 Jul 31;21(1):304. doi: 10.1186/s12876-021-01885-4. PMID 34332533